CLINICAL TRIAL: NCT06141291
Title: Neuromuscular Decline After Physical Inactivity: a Comparison of Younger and Older Adults
Brief Title: Bed Rest Study SBI 2023
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science and Research Centre Koper (Other)
Collaborators: Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI) (Unknown); Izola General Hospital (Other); University of Padova (Other); University of Udine (Other); University of Pavia (Other); University of Trieste (Other)
Responsible Party: Principal Investigator, Rado Pisot, Director, Scientific councillor, Science and Research Centre Koper
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BEDREST
Record Dates: First submitted 2023-10-11; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Healthy Aging; Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Diet, High-Protein; Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Old 1 (Other): 1. Assessment of changes in insulin sensitivity (Oral Glucose Tolerance test and muscle insulin signalling: immunofluorescence and western blot of GLUT-4, IRS-1, MPP/TIMP, etc.) following bed rest in old and young subjects.
  Interventions: Diagnostic Test: OGTT
- Old 2 (Experimental): 1. Assessment of changes in insulin sensitivity (Oral Glucose Tolerance test and muscle insulin signalling: immunofluorescence and western blot of GLUT-4, IRS-1, MPP/TIMP, etc.) following bed rest in old and young subjects.
  2. Test the ability of high protein diet (1.4 g protein/kg/day) with branched chain amino acid and cysteine supplementation to decrease bed rest induced muscle atrophy, glutathione depletion and insulin resistance in old subjects.
  Interventions: Dietary Supplement: High protein diet; Diagnostic Test: OGTT
- Young (Other): 1. Assessment of changes in insulin sensitivity (Oral Glucose Tolerance test and muscle insulin signalling: immunofluorescence and western blot of GLUT-4, IRS-1, MPP/TIMP, etc.) following bed rest in old and young subjects.
  Interventions: Diagnostic Test: OGTT

INTERVENTIONS:
Dietary Supplement: High protein diet — Test the ability of high protein diet (1.4 g protein/kg/day) with branched chain amino acid and cysteine supplementation to decrease bed rest induced muscle atrophy, glutathione depletion and insulin resistance in old subjects.
  Arms: Old 2
Diagnostic Test: OGTT — Assessment of changes in insulin sensitivity (Oral Glucose Tolerance test and muscle insulin signalling: immunofluorescence and western blot of GLUT-4, IRS-1, MPP/TIMP, etc.) following bed rest in old and young subjects.

SUMMARY:
The study will consist of three groups of subjects. Ten young male subjects (18-30 years) will lie supine for 21 days, 10 older male subjects (65+ years) will lie supine for 10 days, and a third group of 10 older male subjects (65+ years) will also lie supine for 10 days but will receive interventions (see below) to counteract the physical changes caused by supine lying. All three groups will be bedridden in the premises of Izola General Hospital. Subjects will be housed in 5-bed rooms at the hospital and will receive 24-hour medical care, proper hygiene, nutrition, passive exercise, Internet, a relaxing environment, and visits. After their stay, subjects return home but receive 21 days of care at local fitness centers. Rehabilitation consists of interval training, in which subjects perform high-intensity exercise for 4 times 5 minutes. A number of important health parameters are measured before, during, and after bed rest. Some of these measurements will be invasive (blood and muscle sampling), for which appropriate medical personnel, sterile instruments, and environment will be available. Measurements will include normal voluntary efforts (indoor cycling, various jumps, short stretches) and electrically evoked muscle contractions (electrical stimulation with single impulses). All tests are normal tests and come from normal lifestyles and routine medical examinations.

ELIGIBILITY:
Inclusion Criteria:

* age: for young arm (18-35), for old arm (65-75)
* BMI: 22 in 32 kg/m2
* appendicular muscle mass > 7,23 kg/m2

Exclusion Criteria:

* serious acute or chronic diseases: skeletal, cancer, cardiovascular, metabolic, neuromuscular and psychiatric;
* cardiovascular disease detected on ECG examination;
* allergies to the active substances used in the study;
* problems with digestion of the active substances;
* frequent diarrhea and vomiting;
* arterial hypertension (>140/90 mmHg);
* psychological problems;
* susceptibility to deep vein thrombosis (D-dimer < 500 μg/L)
* poor orthostatic tolerance (frequent dizziness when changing position, especially when rising from a supine position);
* venous abnormalities that would cause difficulty in drawing blood;
* a large blood volume (more than 300 ml) in the last 3 months prior to the start of the project;
* problems with excessive consumption of alcoholic beverages;
* active smoking;
* Previous participation in any biomedical research in the last 3 months prior to the start of this study;
* a communicable disease before the start of the project;
* any ferromagnetic implant.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 10 days
  Assessment in changes in insulin sensitivity will be made with the use of Oral Glucose Tolerance test (OGTT).

SECONDARY OUTCOMES:
Muscle mass | 10 day
  Muscle mass will be measured with bioimpedance and with DXA.
Muscle force | 10 days
  Quadriceps femoris maximal voluntary contractions (MVC) in isometric conditions at knee angle set at 30 deg flexion and hip fixed at 90 deg flexion using a custom-made knee dynamometer fitted with a load cell (RS 206-0290).
Neuromuscular junction stability | 10 days
  We will evaluate the presence of NMJ stability by analysing: AChR subunits expression

CONTACTS AND LOCATIONS:
Overall Officials: Rado Pišot, PhD, Principal Investigator — Science and Research Centre Koper
Locations (1):
- SRC Koper, Koper, Slovenia

IPD SHARING:
Plan to Share IPD: No